CLINICAL TRIAL: NCT05008484
Title: Effects of Electrical Stimulation and Vitamin D Supplementation on Bone Health Following Spinal Cord Injury
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Virginia Commonwealth University (Other); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B3529-M
Record Dates: First submitted 2021-08-06; First posted 2021-08-17 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury
Keywords: Vitamin D; Electrical Stimulation; Bone Density; Cancellous Bone; Spinal Cord Injury; Rehabilitation; Rowing Exercise
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Methods; Vitamin D; Range of Motion, Articular

STUDY DESIGN:
Intervention Model Description: There are two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NMES Plus Vitamin D (Experimental): Subjects will undergo 4.5 months of open kinematic chain resistance training followed by 4.5 months of closed kinematic chain using simple rowing approach and 2000IU oral vitamin D supplementation daily for 9 months.
  Interventions: Device: NMES; Drug: Vitamin D
- Passive movement plus vitamin D (Active Comparator): Subjects will undergo 9 months of simple passive movement exercise at home and 2000IU oral vitamin D supplementation daily for 9 months.
  Interventions: Drug: Vitamin D; Behavioral: Passive movement

INTERVENTIONS:
Device: NMES — Subjects will undergo 4.5 months of open kinematic chain resistance training followed by 4.5 months of closed kinematic chain using simple rowing approach
  Other Names: Intervention
  Arms: NMES Plus Vitamin D
Drug: Vitamin D — 2000IU oral vitamin D supplementation daily for 9 months
  Other Names: Concomitant therapy
Behavioral: Passive movement — Subjects will perform simple passive movement exercise for their legs while sitting in their wheelchairs at their home. The frequency of the training will be twice weekly
  Other Names: Control
  Arms: Passive movement plus vitamin D

SUMMARY:
Neurogenic osteoporosis is a common complication of spinal cord injury (SCI) that is associated with low impact bone fractures. It is concerning that more than 46,000 Veterans affected with SCI and are at risk of osteoporosis and possible low impact fractures. About fifty percent of all individuals with SCI will develop low impact fracture in their life time. The management of osteoporosis-related fractures can impose substantial economic burden on the health care system, the individual and the families. Previous studies did not succeed in reversing the process of bone loss after SCI. In the present pilot study, we will evaluate the effect of Neuromuscular Electrical Stimulation Resistance Training in combination with oral Vitamin D supplementation, on bone quality in Veterans with chronic SCI, using a randomized experimental design.

DETAILED DESCRIPTION:
Neurogenic osteoporosis is a devastating problem that is likely to impact 46,000 Veterans with chronic spinal cord injury (SCI). It is typically associated with low impact fractures of long bones and other medical comorbidities. It is estimated that approximately fifty percent of all individuals with SCI will develop low impact fracture during their lifetime. The management of osteoporosis related fractures can impose substantial economic burden on the health care system, individuals with SCI and their families. Advancement in medical research clearly indicated that neurogenic osteoporosis is linked to reduced loading and Vitamin D (Vit D) deficiency. Our pilot work indicated that a simple rehabilitation paradigm targeting towards evoking skeletal muscle hypertrophy may attenuate deterioration in trabecular bone parameters after SCI. Evoked resistance training (RT) using surface neuromuscular electrical stimulation (NMES) has been shown as a successful and feasible home-based approach to load skeletal muscles after SCI. Our earlier results may imply long-term compliance and adherence if successfully applied in conjunction with a telehealth approach. In the present study, we propose a simple home-based approach of using NMES RT in conjunction with oral Vit D supplementation on trabecular bone quality in 20 Veterans with chronic SCI. Data will include measurements of trabecular bone quality as determined by magnetic resonance imaging (MRI) and bone biomarkers associated with the process of bone remodeling.

Twenty participants with chronic (> 1-year post-injury) motor complete (AIS A and B) SCI (18 to 65 years of age) will be randomly assigned into either NMES RT plus 2000IU of Vit D (10 participants) or passive movement plus 2000IU Vit D (10 participants) to participate in a repeated measure design trial for 9 months. The NMES RT plus Vit D will undergo 4.5 months of open kinematic chain resistance training followed by 4.5 months of closed kinematic chain using simple rowing approach. This pilot work will have two main specific aims. Aim 1. To determine the impact of home-based NMES RT protocol plus oral Vit D supplementation compared to passive movement plus oral Vit D on bone microarchitectural properties. Aim 2. To determine the impact of home-based NMES RT protocol plus oral Vit D compared to passive movement and Vit D supplementation on biomarkers of bone formation and bone resorption.

ELIGIBILITY:
Inclusion Criteria:

To be included, participants will have to:

* Be 18-65 years of age
* Have history of traumatic SCI ( 1-year) with NLI of C8-T10 and AIS A or B (confirmed by AIS examination performed by PI or a qualified Provider
* Have a caregiver who is available and willing to be trained to apply intervention protocol in the home (placing weights and positioning the Veteran) throughout study duration
* Be a wheelchair user for primary mode of mobility
* Have Knee extensors that must respond to standard surface electrical stimulation procedures (stimulation frequency procedures, 30 Hz; pulse duration:1 ms and amplitude of the current of less than200 mA)
* Be able to receive written clearance from their medical Providers to ensure safety of participants
* Be a Veteran (male or female), however, the Department of Veteran Affairs has limited number of female Veterans, especially those with motor complete injury at level C8-T10 (currently, there are only 3 female Veterans with the target NLI in our SCI registry). Hence, inclusion of women Veterans may be challenging due to this disparity in the SCI population. If we fail to recruit 20 Veterans, we may seek an IRB approval to recruit non-Veterans to meet our target sample size
* Have normal ECG
* Commit to undergo 9 months of trial; 4.5 months of open-kinematic chain resistance training followed by 4.5 months of closed-kinematic chain using simple rowing approach + Vit. D supplementation (Experimental group) or 9 months of passive movement +Vit D supplementation (control group)

Exclusion Criteria:

Potential participants will be excluded if they exhibit any of the following:

* Neurological injury other than SCI
* Older than 65 years of age as they may likely have considerable amount of bone loss at that age
* Have severe osteoporosis because loading porous/fragile bone by electrical stimulation may result in bone fracture
* Those classified as AIS C & D, as they may already be engaging in weight bearing activities that may confound the results of this trial
* Unhealed or unstable fractures in either lower or upper extremities
* Severe scoliosis, deformities in the hip, knee, or ankles OR impaired range-of-motion, as these could be a barrier to safe positioning on the rowing machine, and on MRI or DXA tables
* No caregiver or family member/significant other, willing to help with placing weights and positioning participants' lower extremities on the rowing machine
* Untreated or uncontrolled hypertension (systolic blood pressure (BP) > 140 mmHg; diastolic BP > 90 mmHg), and/or sudden hypotension upon transferring from bed to wheelchair, characterized by a drop in BP by 20 mmHg (especially in persons with tetraplegia) or heart rate > 100 beats per minute
* Anti-coagulation or anti-platelet therapy (including aspirin)
* Implanted pacemakers, implanted defibrillator devices or any metallic implants including knee or hip implants
* Presence of bullets in vertebral column or shrapnel anywhere in the body that may interfere with MRI procedure
* Other medical conditions including cardiovascular disease, uncontrolled type II DM, active deep vein thrombosis (DVT), uncontrolled autonomic dysreflexia, use of insulin for DM management, pressures injuries of stage 3 or higher, or active urinary tract infection
* Severe hypercalcemia (serum calcium > 16mg/dl), stage III-V kidney disease, post-menopausal or estrogen dependent female, and men undergoing anti-androgen therapy or are post orchiectomy
* DXA total body T-score less than -2.5. Total hip BMD T-scores < -3.5 and knee BMD scores of less than 0.6 g/cm2
* Untreatable severe spasticity bearing on potential participants' activities of daily living, such as transfers from bed to wheelchair or maintaining position in wheelchair
* Any psychiatric illness confounding judgment or cognitive impairment in participant or caregiver who is expected to help participant in the trial
* Those with prosthetic lower limbs
* Any condition that, in the judgment of the PI or other medical Providers, preclude safe participation in the study and/or has the potential to expose/increase participant's risk of infection
* Unable to tolerate increasing either electrical stimulation current or weights to the lower legs for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dora E Ifon, PhD, Principal Investigator — Hunter Holmes McGuire VA Medical Center, Richmond, VA
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holman ME, Chang G, Ghatas MP, Saha PK, Zhang X, Khan MR, Sima AP, Adler RA, Gorgey AS. Bone and non-contractile soft tissue changes following open kinetic chain resistance training and testosterone treatment in spinal cord injury: an exploratory study. Osteoporos Int. 2021 Jul;32(7):1321-1332. doi: 10.1007/s00198-020-05778-2. Epub 2021 Jan 14. PMID 33443609
- [Background] Ifon DE, Ghatas MP, Davis JC, Khalil RE, Adler RA, Gorgey AS. Long-term effect of intrathecal baclofen treatment on bone health and body composition after spinal cord injury: A case matched report. World J Orthop. 2020 Oct 18;11(10):453-464. doi: 10.5312/wjo.v11.i10.453. eCollection 2020 Oct 18. PMID 33134108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a spinal cord injury outpatient clinic. One participant was referred by another participant.
Pre-assignment Details: One participant was excluded prior to the start of the study because he failed to complete baseline screening and did not respond to phone calls.
Groups:
- Passive Movement Plus Vitamin D: Subjects will undergo 9 months of simple passive movement exercise at home and 2000IU oral vitamin D supplementation daily for 9 months.
  Vitamin D: 2000IU oral vitamin D supplementation daily for 9 months
  Passive movement: Subjects will perform simple passive movement exercise for their legs while sitting in their wheelchairs at their home. The frequency of the training will be twice weekly. .
Period: Overall Study
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Started | 4 | 2
Completed | 3 (One participant withdrew after the first 4.5 months.) | 1 (One participant withdrew after the first 4.5 months to undergo a surgical procedure not related to the study.)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Six individuals participated in the study. Two participants withdrew after the first phase of the trial (one in the Passive movement plus vitamin D (PM + D), and the other in the NMES + Vit. D group, respectively. As a result, the final number of participants analyzed at 9 months were 4 (3 in the NMES + D group and 1 in the PM + D group).
Groups:
- Total: Total of all reporting groups
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53.5 [45.5 to 54.75] | 42 [35 to 49.5] | 53 [35 to 55.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Trabecular plate width (Tb.PW) in μm as measured by MRI [Median (Inter-Quartile Range); unit: μm] — Trabecular plate width, measured by a trained technician using non-contrast MRI of the femur and tibia with a 3.0T magnet (GE Discovery MR750 software, version: DV24 System 804675VA3T; GE Waukesha, WI). A specific knee coil with a 3D fast-spin gradient echo (10 min) sequence was used to obtain high-resolution images (20-22 FOV). A bilateral phased array coil (USA Instruments) was used to collect 30 contiguous 1-mm slices in the axial plane, starting with the distal end of the femur, and another set of 30 starting with the proximal end of the tibia. Metrics reported as median and IQR.
  μm
    Tb.PW for left femur and tibia | 1791.44 [1760.91 to 1800.50] | 1779.66 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 1791.44 [1759.86 to 1804.14]
    Tb.PW for right femur and tibia | 1769.03 [1729.92 to 1797.23] | 1829.0 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 1789.23 [1755.04 to 1805.46]
Baseline Trabecular spacing (Tb.Sp) (um) as measured by MRI [Median (Inter-Quartile Range); unit: μm] — Trabecular spacing in μm was measured by a non-contrast MRI of the femur and tibia by a trained technician using a 3.0T magnet (GE Discovery MR750 software, version: DV24 System 804675VA3T; GE Waukesha, WI). A specific knee coil with a 3D fast-spin gradient echo (10 min) sequence was used to obtain high-resolution images (20-22 FOV). A bilateral phased array coil (USA Instruments) was used to collect 30 contiguous 1-mm slices in the axial plane, starting with the distal end of the femur, and another set of 30 starting with the proximal end of the tibia. Median and IQR are reported.
  μm
    Tb.Sp for left femur and tibia | 576.16 [489.86 to 665.21] | 430.68 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 486.66 [458.01 to 617.70]
    Tb.Sp for right femur and tibia | 613.71 [520.74 to 720.0] | 445.60 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 509.55 [455.99 to 654.60]
Baseline Trabecular network area density (Tb.NA) (mm^2/mm^3) measured by MRI [Median (Inter-Quartile Range); unit: mm^2/mm^3] — Trabecular network area density (mm^2/mm^3), measured with a non-contrast MRI, of the femur and tibia by a trained technician using a 3.0T magnet (GE Discovery MR750 software, version: DV24 System 804675VA3T; GE Waukesha, WI). A specific knee coil with a 3D fast-spin gradient echo (10 min) sequence was used to obtain high-resolution images (20-22 FOV). A bilateral phased array coil (USA Instruments) was used to collect 30 contiguous 1-mm slices in the axial plane, starting with the distal end of the femur, and another set of 30 starting with the proximal end of the tibia; median and IQR.
  mm^2/mm^3
    Tb.NA for left femur and tibia | 0.44 [0.39 to 0.50] | 0.61 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 0.51 [0.42 to 0.55]
    Tb.NA for right femur and tibia | 0.42 [0.38 to 0.49] | 445.60 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 0.51 [0.40 to 0.56]
Baseline Distal Femur Bone Mineral Density (BMD) in g/cm2 as measured by DXA [Median (Inter-Quartile Range); unit: g/cm2] — A dual-energy X-ray absorptiometry scan was performed by a trained technologist using a General Electric iDXA scanner (GE Lunar Inc., Madison, WI) at baseline, 4.5 months, and at 9 months. The scanner was calibrated using a phantom calibration box that mimics human tissues to assess scan precision and reliability. All participants had their jewelry removed before being placed supine on the scanning table with their arms internally rotated and palms facing medially. Participants received scans in the region of interest on both sides (L & R) of the body (hip, knee), as well as the lumbar spine.
  g/cm2
    Left distal femur BMD | 0.96 [0.83 to 1.15] | 1.20 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 1.12 [0.90 to 1.23]
    Right distal femur BMD | 0.96 [0.82 to 1.13] | 1.22 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 1.10 [0.89 to 1.25]
Baseline Proximal tibia Bone Mineral Density in g/cm2 as measured by DXA. [Median (Inter-Quartile Range); unit: g/cm2] — A dual-energy X-ray absorptiometry scan was performed by a trained technologist using a General Electric iDXA scanner (GE Lunar Inc., Madison, WI) at baseline, 4.5 months, and at 9 months. The scanner was calibrated using a phantom calibration box that mimics human tissues to assess scan precision and reliability. All participants had their jewelry removed before being placed supine on the scanning table with their arms internally rotated and palms facing medially. Participants received scans in the region of interest on both sides (L & R) of the body (hip, knee), as well as the lumbar spine.
  g/cm2
    Left proximal tibia BMD | 0.97 [0.95 to 1.09] | 1.50 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 1.19 [0.96 to 1.40]
    Right proximal tibia BMD | 1.0 [0.91 to 1.13] | 1.5 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 1.20 [0.97 to 1.36]
Baseline Bone formation marker (Procollagen Type 1 Intact N-Propeptide [P1NP] in mcg/L [Median (Inter-Quartile Range); unit: mcg/L] — Fasting blood samples were obtained by venopuncture by the same person at approximately the same time of day and under similar conditions to assess P1NP, a marker of bone formation. Specimens were analyzed by Quest Diagnostics (Nichols Institute, Chantilly, VA). The reference range for PINP is 30-110 mcg/L, and an increase denotes poor bone health.
  mcg/L | 39 [35.5 to 67.75] | 63.5 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 46 [26 to 82]
Baseline Bone resorption marker (C-telopeptide of Type I collagen [CTX]), in pg/mL [Median (Inter-Quartile Range); unit: pg/mL] — CTX is a biochemical marker of bone resorption. Fasting blood samples were obtained from participants with venopuncture by the same person at approximately the same time of day and under similar conditions to measure CTX (pg/mL). Specimens were analyzed by Quest Diagnostics (Nichols Institute, Chantilly, VA). Sex and age-related reference ranges for males: 18-29yrs (87-1200), 30-39yrs (70-780), 40-49yrs (60-700), and 50-68yrs (87-345). CTX is released into the circulation when osteoclasts degrade bone matrix; thus, higher levels reflect increased osteoclastic activity and faster bone turnover.
  pg/mL | 351.5 [284.25 to 506.25] | 531 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 418 [285 to 638]
Baseline Serum concentration of 25-hydroxyvitamin D in ng/mL [Median (Inter-Quartile Range); unit: ng/mL] — 25 (OH)D is the main circulating form of vit. D, and the most reliable biochemical marker of an individual's vitamin D status. It is crucial for maintaining bone strength, mineral balance, and overall bone health. Adequate levels of 25(OH)D improve intestinal calcium absorption, which is vital for normal bone formation and remodeling. Low levels lead to decreased calcium absorption, resulting in secondary hyperparathyroidism, which in turn leads to increased bone resorption and weakening of the bone structure. Normal range is 32 to 100; < 20 ng/mL is deficiency, and 20 to 29 is insufficiency.
  ng/mL | 23.4 [17.9 to 29.25] | 26.05 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 25.3 [19.05 to 29.83]
Baseline Physical domain of Quality of life measure [Median (Inter-Quartile Range); unit: units on a scale (0-100)] — The WHOQOL-BREF, a 26-item self-administered questionnaire, assesses quality of life across four domains, including two general items. Each item is rated on a 5-point Likert scale (1 = negative or low perception, 5 = positive or high perception). Physical health (7 items) evaluates energy, fatigue, sleep, mobility, pain, and activities of daily living. The maximum score for this domain is 100, and a higher score indicates better physical health.
  units on a scale (0-100) | 72 [62.75 to 78.25] | 75 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 72 [69 to 79.5]
Baseline Psychological health domain of Quality of life measure [Median (Inter-Quartile Range); unit: units on a scale (0-100)] — The WHOQOL-BREF, a 26-item self-administered questionnaire, assesses quality of life across four domains, including two general items. Each item is rated on a 5-point Likert scale (1 = negative or low perception, 5 = positive or high perception). Psychological health (6 items) measures self-esteem, body image, negative and positive feelings, and concentration. The maximum score for this domain is 100, and a higher score indicates better psychological health.
  units on a scale (0-100) | 65.5 [48.5 to 84.25] | 81 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 81 [57.75 to 81]
Baseline Social relationship domain of Quality of life measure. [Median (Inter-Quartile Range); unit: units on a scale (0-100)] — The WHOQOL-BREF, a 26-item self-administered questionnaire, assesses quality of life across four domains, including two general items. Each item is rated on a 5-point Likert scale (1 = negative or low perception, 5 = positive or high perception). Social relationships (3 items) assess personal relationships, social support, and sexual life. The maximum score for this domain is 100, and a higher score indicates a better quality of life in the social relationships domain.
  units on a scale (0-100) | 75 [64.25 to 84.25] | 78 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 78 [70.5 to 81]
Baseline environmental engagement domain of Quality of life measure. [Median (Inter-Quartile Range); unit: units on a scale (0-100)] — The WHO Quality of Life (WHOQOL)-BREF, a 26-item self-administered questionnaire, assesses quality of life across four domains, including two general items. Each item is rated on a 5-point Likert scale (1 = negative or low perception, 5 = positive or high perception). Environmental engagement (8 items) assesses financial resources, safety, home environment, health care access, and opportunities for recreation and learning. The maximum score for this domain is 100, and a higher score indicates a better quality of life in the environmental domain.
  units on a scale (0-100) | 84.5 [79.5 to 89.5] | 81 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm. | 81 [81 to 86.25]

OUTCOME MEASURES:

1. Primary Outcome: Change in Trabecular Plate Width (Tb.PW) for Femur and Tibia at 4.5 Months
Description: The outcome measure was trabecular plate width expressed in μm, as measured by a non-contrast magnetic resonance imaging (MRI) of the femur and tibia. A trained radiology technician performed the MRI using a 3.0T magnet (GE Discovery MR750 software, version: DV24 System 804675VA3T; GE Waukesha, WI). A specific knee coil with a 3D fast-spin gradient echo (10 min) sequence was used to obtain high-resolution images (20-22 FOV). A bilateral phased array coil (USA Instruments) was used to collect 30 contiguous 1-mm slices in the axial plane, starting with the distal end of the femur, and another block of 30 starting with the proximal end of the tibia. The metric used was the median change from baseline to 4.5 months and 9 months, respectively. Higher values indicate improved bone trabeculae.
Time Frame: 4.5 months
Population: Participants (n = 6) with chronic motor-complete spinal cord injury (C8-T10) with ASIA impairment classification of A or B, completed an MRI at baseline and 4.5 months.
Measure: Median (Inter-Quartile Range); unit: μm
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 4 | 2
μm
  Left Femur and TibiaTb.PW at 4.5 months | 1785.42 [1753.76 to 1809.26] | 1819.41 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm.
  Right Femur and Tibia Tb.PW at 4.5 months | 1805.52 [1773.62 to 1816.2] | 1834.67 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm.

2. Primary Outcome: Change in Trabecular Plate Width (Tb.PW) for Femur and Tibia at 9 Months
Description: The outcome measure was trabecular spacing expressed in μm, as measured by a non-contrast magnetic resonance imaging (MRI) of the femur and tibia. A trained radiology technician performed the MRI using a 3.0T magnet (GE Discovery MR750 software, version: DV24 System 804675VA3T; GE Waukesha, WI). A specific knee coil with a 3D fast-spin gradient echo (10 min) sequence was used to obtain high-resolution images (20-22 FOV). A bilateral phased array coil (USA Instruments) was used to collect 30 contiguous 1-mm slices in the axial plane, starting with the distal end of the femur, and another set of 30 slices starting with the proximal end of the tibia. The metric used was the median change from baseline to 9 months. Higher values indicate improved Tb. PW.
Time Frame: 9 months
Population: Four participants with chronic motor-complete spinal cord injury (C8-T10) and an ASIA impairment classification of A or B completed MRI at 9 months (n = 3 in the NMES + Vit. D group and n = 1 in the Passive movement + Vit. D group).
Measure: Median (Inter-Quartile Range); unit: um
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
um
  Left Femur and Tibia Tb.PW at 9 months | 1767.38 [1762.70 to 1779.56] | 1750.77 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.
  Right Femur and Tibia Tb.PW at 9 months | 1786.44 [1775.62 to 1796.93] | 1734.01 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.

3. Primary Outcome: Change in Trabecular Spacing (Tb.Sp) for Femur and Tibia at 4.5 Months
Description: The outcome measure was trabecular spacing expressed in μm, as measured by a non-contrast magnetic resonance imaging (MRI) of the femur and tibia. The metric used was the median change from baseline to 4.5 months and 9 months, respectively. Higher values indicate poorer bone health. A trained radiology technician performed the MRI using a 3.0T magnet (GE Discovery MR750 software, version: DV24 System 804675VA3T; GE Waukesha, WI). A specific knee coil with a 3D fast-spin gradient echo (10 min) sequence was used to obtain high-resolution images (20-22 FOV). A bilateral phased array coil (USA Instruments) was used to collect 30 contiguous 1-mm slices in the axial plane, starting with the distal end of the femur, and another block of 30 starting with the proximal end of the tibia.
Time Frame: 4.5 months
Population: Six participants with chronic motor-complete spinal cord injury (C8-T10) and ASIA impairment classification of A or B completed MRI at 4.5 months (n = 4 in the NMES + Vit. D group and n = 2 in the Passive movement + Vit. D group).
Measure: Median (Inter-Quartile Range); unit: um
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 4 | 2
um
  Left femur and tibia Tb.Sp at 4.5 months | 550.41 [523.63 to 583.66] | 463.22 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.
  Right femur and tibia Tb.Sp at 4.5 months | 556.84 [532.04 to 588.58] | 440.57 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.

4. Primary Outcome: Change in Trabecular Spacing (Tb.Sp) for Femur and Tibia at 9 Months
Description: The outcome measure was trabecular plate width expressed in μm, as measured by a non-contrast magnetic resonance imaging (MRI) of the femur and tibia. A trained radiology technician performed the MRI using a 3.0T magnet (GE Discovery MR750 software, version: DV24 System 804675VA3T; GE Waukesha, WI). A specific knee coil with a 3D fast-spin gradient echo (10 min) sequence was used to obtain high-resolution images (20-22 FOV). A bilateral phased array coil (USA Instruments) was used to collect 30 contiguous 1-mm slices in the axial plane, starting with the distal end of the femur, and another block of 30 beginning with the proximal end of the tibia. The metric used was the median change from baseline to 4.5 months and 9 months, respectively. Higher values indicate improved bone trabeculae.
Time Frame: 9 months
Population: Four participants with motor complete spinal cord injury (C8-T10) ( 3 in the NMES + vit DArm and 1 in the Passive movement + Vit.D Arm) underwent MRI at 9 months.
Measure: Median (Inter-Quartile Range); unit: um
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
um
  Left femur and tibia Tb.Sp at 9 months | 494.33 [493.58 to 503.24] | 526.39 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.
  Right femur and tibia Tb.Sp at 9 months | 484.05 [482.67 to 518.45] | 565.33 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm,

5. Primary Outcome: Change in Trabecular Network Area Density (Tb.NA) Measured in mm^2/mm^3) at 4.5 Months
Description: The outcome measure was trabecular network area density expressed in mm^2/mm^3, as measured by a non-contrast magnetic resonance imaging (MRI) of the femur and tibia. The metric used was the median change from baseline to 4.5 months and 9 months, respectively. Higher values indicate improved bone trabeculae network area density. A trained radiology technician performed the MRI using a 3.0T magnet (GE Discovery MR750 software, version: DV24 System 804675VA3T; GE Waukesha, WI). A specific knee coil with a 3D fast-spin gradient echo (10 min) sequence was used to obtain high-resolution images (20-22 FOV). A bilateral phased array coil (USA Instruments) was used to collect 30 contiguous 1-mm slices in the axial plane, starting with the distal end of the femur, and another block of 30 starting with the proximal end of the tibia.
Time Frame: 4.5 months
Population: All participants (n = 6) with chronic motor-complete spinal cord injury (C8-T10) and ASIA impairment classification of A or B completed an MRI at baseline and at 4.5 months. By 9 months, only four participants (n = 3 in the NMES + Vit. D group and n = 1 in the Passive movement + Vit. D group) completed the MRI after two participants (one in each group) voluntarily withdrew.
Measure: Median (Inter-Quartile Range); unit: mm^2/mm^3
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 4 | 2
mm^2/mm^3
  Left femur and tibia Tb.NA at 4.5 months | 0.48 [0.44 to 0.54] | 0.59 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm.
  Right femur and tibiaTb.NA at 4.5 months | 0.45 [0.44 to 0.48] | 0.46 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm.

6. Primary Outcome: Change in Trabecular Network Area Density (Tb.NA) as Measured by MRI at 9 Months
Description: as for outcome 5
Time Frame: 9 months
Population: Four participants with motor complete spinal cord injury (C8-T10), underwent MRI of both knees upon completion of the trial.
Measure: Median (Inter-Quartile Range); unit: mm^2/mm^3
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
mm^2/mm^3
  Left femur and tibia Tb.NA at 9 months | 0.52 [0.52 to 0.54] | 0.48 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.
  Right femur and tibia Tb.NA at 9 months | 0.54 [0.53 to 0.55] | 0.44 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.

7. Secondary Outcome: Change in Bone Mineral Density in Distal Femur as Measured by Dual Energy X-ray Absorptiometry (DXA) Scan
Description: A dual-energy X-ray absorptiometry scan was performed by a trained technologist using a General Electric iDXA scanner (GE Lunar Inc., Madison, WI) at baseline, 4.5 months, and at 9 months. The scanner was calibrated using a phantom calibration box that mimics human tissues to assess scan precision and reliability. All participants had their jewelry removed before being placed supine on the scanning table with their arms internally rotated and palms facing medially. Participants received scans in the region of interest on both sides (L & R) of the body (hip, knee), as well as the lumbar spine.
Time Frame: 4.5 months
Population: Six males with motor complete spinal cord injury (C8-T10) underwent DXA scans after 4.5 months in the trial.
Measure: Median (Inter-Quartile Range); unit: g/cm2
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 4 | 2
g/cm2
  Left distal femur BMD | 0.94 [0.85 to 1.08] | 1.17 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this study Arm.
  Right distal femur BMD | 0.90 [0.81 to 1.04] | 1.21 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this study Arm.
Statistical Analysis 1: Comparison: NMES Plus Vitamin D vs Passive Movement Plus Vitamin D; Test type: Superiority

8. Secondary Outcome: Change in Distal Femur Bone Mineral Density
Description: as for outcome 7
Time Frame: 9 months
Population: Four males with motor complete spinal cord injury (C8-T10) underwent DXA scans upon completing the trial.
Measure: Median (Inter-Quartile Range); unit: g/cm2
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
g/cm2
  Left distal femur BMD | 0.84 [0.81 to 1.0] | 1.07 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.
  Right distal femur BMD | 0.84 [0.78 to 0.96] | 1.02 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.

9. Secondary Outcome: Change in Proximal Tibia Bone Mineral Density (BMD) as Measured by Dual-energy X-ray Absorptiometry (DXA) Scan
Description: as for outcome 7
Time Frame: 4.5 months
Population: Four males with motor complete spinal cord injury (C1-T10) underwent DXA of the knees after 4.5 months of the trial.
Measure: Median (Inter-Quartile Range); unit: gm/cm2
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 4 | 2
gm/cm2
  Left proximal tibia BMD | 0.97 [0.92 to 1.06] | 1.47 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm.
  Right proximal tibia BMD | 1.09 [0.93 to 1.24] | 1.42 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm.

10. Secondary Outcome: Change in Proximal Tibia Bone Mineral Density as Measured by a Dual-energy X-ray Absorptiometry (DXA) Scan
Description: as for outcome 7
Time Frame: 9 months
Population: Four males with motor complete spinal cord injury (C8-T10) underwent DXA scan of the knees after 9 months of the trial.
Measure: Median (Inter-Quartile Range); unit: gm/cm2
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
gm/cm2
  Left proximal tibia BMD | 1.02 [0.98 to 1.03] | 1.3 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.
  Right proximal tibia BMD | 1.09 [0.97 to 1.18] | 1.24 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.

11. Secondary Outcome: Change in Bone Formation Marker - Procollagen Type 1 N-terminal Propeptide (P1NP) in mcg/L
Description: Fasting blood samples were collected by venipuncture by the same individual at roughly the same time of day and under similar conditions to evaluate P1NP, a marker of bone formation. Samples were analyzed at Quest Diagnostics (Nichols Institute, Chantilly, VA). The reference range for P1NP is 30-110 mcg/L, and an increase indicates poor bone health.
Time Frame: 4.5 months
Population: Six males with motor complete spinal cord injury (C8-T10).
Measure: Median (Inter-Quartile Range); unit: mcg/L
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 4 | 2
mcg/L | 38 [35 to 45] | 53 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm.

12. Secondary Outcome: Change in Bone Formation Marker - Procollagen Type 1 Intact N-Propeptide (P1NP) Measured in mcg/L
Description: as for outcome 11
Time Frame: 9 months
Population: Four males with motor complete spinal cord injury (C8-T10)
Measure: Median (Inter-Quartile Range); unit: mcg/L
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
mcg/L | 35 [34 to 38.5] | 34 [NA to NA] — IQR values could not be calculated due to only one participant assessed within this Arm.

13. Secondary Outcome: Change in Bone Resorption Marker-C-telopeptide of Type I Collagen (CTX)
Description: CTX is a biochemical marker of bone resorption. Fasting blood samples were collected from participants via venipuncture by the same person at approximately the same time of day and under similar conditions to measure CTX (pg/mL). The samples were analyzed by Quest Diagnostics (Nichols Institute, Chantilly, VA). Sex and age-related reference ranges for males are: 18-29 years (87-1200), 30-39 years (70-780), 40-49 years (60-700), and 50-68 years (87-345). CTX is released into circulation when osteoclasts break down bone matrix; therefore, higher levels indicate increased osteoclastic activity and faster bone turnover.
Time Frame: 4.5 months
Population: Six males with motor complete spinal cord injury (C8-T10)
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 4 | 2
pg/mL | 291 [252.5 to 393.75] | 512.5 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm.

14. Secondary Outcome: Change in Bone Resorption Marker-C-telopeptide of Type I Collagen (CTX)
Description: CTX is a biochemical marker of bone resorption. Fasting blood samples were collected from participants via venipuncture by the same person at approximately the same time of day and under similar conditions to measure CTX (pg/mL). The samples were analyzed by Quest Diagnostics (Nichols Institute, Chantilly, VA). Sex and age-related reference ranges for males are as follows: 18-29 years (87-1200), 30-39 years (70-780), 40-49 years (60-700), and 50-68 years (87-345). CTX is released into circulation when osteoclasts break down bone matrix; therefore, higher levels indicate increased osteoclastic activity and faster bone turnover.
Time Frame: 9 months
Population: Four males with motor complete spinal cord injury (C8-T10).
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
pg/mL | 333 [294 to 367.5] | 306 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.

15. Secondary Outcome: Change in Serum 25-hydroxyvitamin D [25(OD)D] Level
Description: 25-hydroxyvitamin D is the major circulating form of vitamin D and the most reliable biochemical indicator of an individual's vitamin D status.
  It is essential for maintaining bone strength, balance of minerals, and overall bone integrity. Adequate levels of 25(OH)D enhance intestinal calcium absorption for normal bone formation and remodeling. When vitamin D levels are low, calcium absorption decreases, leading to secondary hyperparathyroidism, which in turn increases bone resorption and weakens bone structure. The normal range is 32 to 100 ng/mL. Less than 20ng/mL is considered a deficiency, and 20 to 29 ng/mL is insufficiency.
Time Frame: 4.5 months
Population: Six males with motor complete spinal cord injury (C8-T10).
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 4 | 2
ng/mL | 32.1 [29.2 to 38.08] | 37.15 [NA to NA] — IQR values could not be calculated due to only 2 participants assessed within this Arm.

16. Secondary Outcome: Change in Serum 25-hydroxyvitamin D Level
Description: 25-hydroxyvitamin D is the main circulating form of vitamin D and the most reliable biochemical marker of an individual's vitamin D status. Vitamin D is crucial for maintaining bone strength, mineral balance, and overall bone health. Adequate levels of 25(OH)D improve intestinal calcium absorption, which is vital for normal bone formation and remodeling. When vitamin D levels are low, calcium absorption drops, leading to secondary hyperparathyroidism, which then increases bone resorption and weakens bone structure. The normal range is 32 to 100 ng/mL. Less than 20 ng/mL is considered a deficiency, and 20 to 29 ng/mL indicates insufficiency.
Time Frame: 9 months
Population: Four males with motor complete spinal cord injury (C8 to T10)
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
ng/mL | 49.4 [33.2 to 49.65] | 50.7 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.

17. Secondary Outcome: Change in Quality-of-life Measure: Physical Health (Scored on 1-5 Likert Scale)
Description: The secondary outcome measure was the WHO Quality of Life (WHOQOL)-BREF, a 26-item self-administered questionnaire developed by WHO to assess quality of life across four domains, including two general items. Each item is rated on a 5-point Likert scale (1 = negative or low perception, 5 = positive or high perception). The instrument includes four health domains: physical health, psychological health, social relationships, and environmental engagement. Physical health (7 items) evaluates energy, fatigue, sleep, mobility, pain, and activities of daily living. The maximum score for this domain is 100, and a higher score indicates a better quality of life.
Time Frame: 9 months
Population: Four males with chronic motor-complete spinal cord injury (C8-T10).
Measure: Median (Inter-Quartile Range); unit: units on a scale (0-100)
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
units on a scale (0-100) | 75 [65.5 to 78] | 69 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.
Statistical Analysis 1: Comparison: NMES Plus Vitamin D; Test type: Superiority; Mean Difference (Final Values) = -8, 95% CI 2-sided [-36.6 to 24.6], Standard Error of Mean 11.0

18. Secondary Outcome: Change in Quality-of-life Measure- Psychological Health
Description: The WHOQOL-BREF instrument was used to assess QOL in four domains of health, including: physical health, psychological health, social relationships, and environmental engagement. The mean scores of items within each domain were used to calculate domain scores, which were then transformed using the WHOQOL-BREF scoring manual to make the domain scores comparable to those used in the WHOQOL-100. Items 3, 4, and 26 were reverse-coded per the instruction manual. Psychological health (6 items) measures self-esteem, body image, negative and positive feelings, and concentration. A higher score denotes higher psychological health.
Time Frame: 9 months
Population: Six males with motor-complete spinal cord injury (C8-T10)
Measure: Median (Inter-Quartile Range); unit: score on a scale (0-100)
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
score on a scale (0-100) | 81 [68.5 to 84.5] | 81 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.
Statistical Analysis 1: Comparison: NMES Plus Vitamin D vs Passive Movement Plus Vitamin D; Test type: Superiority; Mean Difference (Final Values) = -13.75, 95% CI 2-sided [-52.1 to 24.6], Standard Error of Mean 12.1

19. Secondary Outcome: Change in Quality-of-life Measure- Social Relationships Domain
Description: The WHOQOL-BREF instrument was used to assess QOL in four domains of health, including: physical health, psychological health, social relationships, and environment. The mean scores of items within each domain were used to calculate domain scores, which were then transformed using the WHOQOL-BREF scoring manual to make the domain scores comparable to those used in the WHOQOL-100. Items 3, 4, and 26 were reverse-coded per the instruction manual. Social relationships (3 items) assess personal relationships, social support, and sexual life. A higher score denotes a higher social relationships.
Time Frame: 9 months
Population: Six males with motor-complete spinal cord injury (C8-T10).
Measure: Median (Inter-Quartile Range); unit: score on a scale (0-100)
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
score on a scale (0-100) | 69 [62.5 to 72] | 75 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.
Statistical Analysis 1: Comparison: NMES Plus Vitamin D vs Passive Movement Plus Vitamin D; Test type: Superiority; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-31.8 to 22.8], Standard Error of Mean 9.8

20. Secondary Outcome: Change in Quality-of-life Measure-environmental Engagement Domain
Description: The WHOQOL-BREF instrument was used to assess QOL in four domains of health participants, including: physical health, psychological health, social relationships, and environmental engagement. The mean scores of items within each domain were used to calculate domain scores, which were then transformed using the WHOQOL-BREF scoring manual to make the domain scores comparable to those used in the WHOQOL-100. Items 3, 4, and 26 were reverse-coded per the instruction manual. Environmental engagement (8 items) assesses financial resources, safety, home environment, health care access, and opportunities for recreation and learning. A Higher score denotes better environmental engagement.
Time Frame: 9 months
Population: Four males with motor complete spinal cord injury (C8 to T10).
Measure: Median (Inter-Quartile Range); unit: units on a scale (0-100)
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
Number analyzed (Participants) | 3 | 1
units on a scale (0-100) | 75 [72 to 78] | 75 [NA to NA] — IQR values could not be calculated due to only 1 participant assessed within this Arm.

ADVERSE EVENTS:
Time Frame: Four weeks. This was a spontaneous reporting by the participant. The participant was followed and monitored by his SCI provider over the 4 weeks period, while research staff maintained weekly contact for updates on participant's healing process.
Description: One participant in the intervention group reported opening of an old ischial wound scar (grade II) due sitting longer than usual on a commode for routine bowel care program.
Arm/Group | NMES Plus Vitamin D | Passive Movement Plus Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 1/4 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NMES Plus Vitamin D (N=4) | Passive Movement Plus Vitamin D (N=2)
Disruption in skin integrity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — One participant reported opening of an ischial wound scar (grade II) due to sitting for a prolonged period of time on a commode to do his bowel care.

LIMITATIONS AND CAVEATS:
The small sample size, only male participants, and a wide variation in participants' level of injury (C8-T10) and age, limit generalizability of the study findings to a broader spinal cord injury population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT05008484/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT05008484/ICF_000.pdf